CLINICAL TRIAL: NCT04101045
Title: Pathogenesis of the Cardiometabolic Risk in Youth With Type 1 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: During the pandemic the funding agency stopped funding studies.
Sponsor: Yale University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000025170
Record Dates: First submitted 2019-09-17; First posted 2019-09-24 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Type 1 Diabetes; De Novo Lipogenesis
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Poorly-controlled T1D (Active Comparator): Patients in this group will have poorly-controlled T1D (HbA1c >8.5%).
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test
- Controlled T1D (Active Comparator): Patients in this group will have T1D and achieve targeted glycemic control (HbA1c <7.5%).
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test
- Lean controls (Active Comparator): Patients in this group will not have T1D.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance Test — Each participant consumes a dinner scaled to his/her energy needs which is prepared by the metabolic kitchen. Dinner will be provided beforehand if patient does this portion at home. The participant consumes the first of three doses of D2O. Two additional doses of D20 are given at on day 1 and on day 2. The total D2O given (3 ml per kg of body water) is designed to raise body deuterium levels to 0.3% and is administered as described above to maintain steady state until the end of the study. At the HRU, an IV catheter will be inserted in order to collect blood to assess DNL. Blood draws begin during the fasting state to assess basal rates of DNL and then for six hours after the consumption of a glucose/fructose beverage (75g glucose and 25g fructose ) to assess postprandial rates of DNL. Blood draws will be taken 15 minutes before ingestion of the sugar beverage, then for every half hour for 6 hours.

SUMMARY:
The purpose of this study is to quantitate hepatic de novo lipogenesis (DNL) in youth with poorly-controlled type 1 diabetes (T1D) (HbA1c >8.5%), youth with T1D who achieve targeted glycemic control (HbA1c <7.5%) and lean controls. Hypothesis: Youth with poor glycemic control experience higher fractional hepatic DNL during the fasting and the postprandial states than youth who achieve targeted glycemic control and lean controls.

DETAILED DESCRIPTION:
What is not known, is whether hepatic de novo lipogenesis (DNL) contributes to dyslipidemia in this in patients with type 1 diabetes (T1D). The aim of the study is to test the hypothesis that an enhanced rate of DNL largely contributes to dyslipidemia occurring in youth with poorly-controlled T1D. According to this hypothesis, youth with poorly-regulated T1D experience a state of persistent insulin independent, highly variable fluctuations of glucose, and other sugars, through the glycolytic pathway that result in an enhancement of hepatic DNL and an increased production of triglycerides (TG). Newly-formed TG are packaged into large-VLDL that are secreted into the circulation contributing to an increase in plasma TG. When the TG concentration in the hepatocytes exceeds the ability of the liver to secrete TG, the latter start accumulating leading to hepatic steatosis.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c >8.5% for the group with poorly controlled diabetes
* HbA1c <7.5% for the well-controlled patients
* T1D for at least 12 months (T1D groups only)
* Negative pregnancy test (all groups)

Exclusion Criteria:

* Baseline creatinine >1
* Being on medications affecting glucose concentrations other than insulin
* Positive pregnancy test
* Endocrinopathies

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Fractional hepatic DNL | Baseline to Six hours
  % Fractional hepatic DNL

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Santoro, MD, PhD, Principal Investigator — Assistant Professor of Pediatrics (Endocrinology)
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monga Kravetz A, Testerman T, Galuppo B, Graf J, Pierpont B, Siebel S, Feinn R, Santoro N. Effect of Gut Microbiota and PNPLA3 rs738409 Variant on Nonalcoholic Fatty Liver Disease (NAFLD) in Obese Youth. J Clin Endocrinol Metab. 2020 Oct 1;105(10):e3575-85. doi: 10.1210/clinem/dgaa382. PMID 32561908